CLINICAL TRIAL: NCT02945072
Title: Postoperative Behavior in Children: A Comparison of Inhalation Anesthesia (Sevoflurane) Versus Total Intravenous Anesthesia (TIVA)
Brief Title: Clinical Study of Behavior Problems in Children After Different Anesthesia Methods
Acronym: PST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Children's Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: KEK-ZH-Nr. 2011-0009
Record Dates: First submitted 2016-10-13; First posted 2016-10-26 (Estimated); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Child Behavior; Problem Behavior
Keywords: Child Behavior; Problem Behavior; postoperative behaviour problems
MeSH Terms: conditions — Child Behavior; Problem Behavior | interventions — Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sevoflurane group (Active Comparator): general anesthesia will be maintained with sevoflurane
  Interventions: Procedure: Sevoflurane
- TIVA group (Experimental): general anesthesia will be maintained with total intravenous anesthesia (propofol and remifentanyl)
  Interventions: Procedure: TIVA

INTERVENTIONS:
Procedure: TIVA — TIVA is use to anesthesia maintenance after anesthesia induction (Propofol 10mg/kg/h, Remifentanil 0.2mcg/kg/min, dose adaptation as required for sufficient anesthesia)
  Arms: TIVA group
Procedure: Sevoflurane — Sevoflurane is use to anesthesia maintenance after anesthesia induction (target et 2 Vol% in 50-70% N2O, dose adaptation as required)
  Arms: Sevoflurane group

SUMMARY:
The aim of this study is to investigate long-lasting or later behavioral changes in children in the context of different anesthesia techniques (Inhalation anesthesia vs. TIVA)

DETAILED DESCRIPTION:
The process of surgery and anaesthesia can be an extremely frightening and stressful event for a child, and is frequently followed by negative postoperative behavioural changes. This Event could be associated with poor postoperative outcome and long term behavior problems like anxiety, eating or sleeping disorders. The aim of this study is to investigate long-lasting or later behavioral changes in children in the context of different anesthesia techniques (Inhalation anesthesia vs. TIVA). After anesthesia initiation, anesthesia maintenance should be done with sevoflurane or Tiva. The effect of behavioral changes in children in the context of anesthesia techniques should be evaluate by post hospitalisation behavior and Strengths and Difficulties Questionnaire at first, second and fourth week. Early postoperative problems like postoperative nausea and vomiting, pain level, pain therapy and postoperative awareness should be evaluate too.

ELIGIBILITY:
Inclusion Criteria:

* elective Operation
* operation in general anesthesia in combination with regional anesthesia
* Age 2-10 years
* ASA classification 1 or 2 (without severe basic disease or disability)

Exclusion Criteria:

* Lack of Consensus
* general anesthesia during the last 3 months before or 4 weeks after the procedure
* PONV prophylaxis with droperidol
* severe known growth factor
* mental pre-existing conditions and behavioral abnormalities
* contraindications for one of the used study medications
* insufficient regional anesthesia
* secondary intervention within of the 4-week follow-up

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 500 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Post-Hospital Behaviour Questionnaire (PHBQ) score postoperatively | first week postoperative
  child's PHBQ score first week postoperatively
Post-Hospital Behaviour Questionnaire (PHBQ) score postoperatively | second week postoperative
  child's PHBQ score second week postoperatively
Post-Hospital Behaviour Questionnaire (PHBQ) score postoperatively | fourth week postoperative
  child's PHBQ score fourth week postoperatively
SDQ Questionnaire score postoperatively | first week postoperative
  child's SDQ score first week postoperatively
SDQ Questionnaire score postoperatively | second week postoperative
  child's SDQ score second week postoperatively
SDQ Questionnaire score postoperatively | fourth week postoperative
  child's SDQ score fourth week postoperatively

SECONDARY OUTCOMES:
postoperative pain Level (by VAS) | in the first postoperative week (3 times a day)
  Visual Analog Scale for Pain (VAS Pain) were used to evaluate postoperative pain level
postoperative pain Level (by CHEOPS) | in the first postoperative week (3 times a day)
  CHEOPS (Children's Hospital of Eastern Ontario Pain Scale) were used to evaluate postoperative pain level
postoperative pain medication | in the first postoperative week
  All pain medications are recorded during the first postoperative week.Nurses and parents recorded all substance and application times by questionnaire.
Intraoperative awareness | in the first and second postoperative day
  In order to record an intraoperative awareness, a semistructured interview is conducted with test questions.
postoperative Nausea and vomiting | in the first and second postoperative day
  Nausea and Vomiting are recognized in frequency and time using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Buehler, MD, Study Chair — University children hosptial Zurich
Locations (1):
- Dr. Philipp Buehler, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No